CLINICAL TRIAL: NCT03850912
Title: SIMPRO Research Center: Integration and Implementation of PROs for Symptom Management in Oncology Practice
Brief Title: Symptom Management Implementation of Patient Reported Outcomes in Oncology
Acronym: SIMPRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); RTI International (Other); Baptist Memorial Health Care Corporation (Other); Dartmouth-Hitchcock Medical Center (Other); MaineHealth (Other); West Virginia University (Other); Lifespan (Other)
Responsible Party: Principal Investigator, Michael Hassett, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 18-734; 1UM1CA233080-01 (NIH)
Record Dates: First submitted 2019-02-20; First posted 2019-02-22 (Actual); Results first posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Other Cancer; Gastrointestinal Cancer; Thoracic Cancer; Gynecologic Cancer
Keywords: Other Cancer; Digital health; Patient reported outcomes; Symptom management
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Intervention Model Description: The primary study design is a hybrid effectiveness-implementation stepped-wedge cluster randomized trial involving several different research activities to assess outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Stakeholder Feedback (Control Period) (Other): Eligible stakeholders at each SIMPRO site were invited to provide feedback through focus groups, team meetings, and surveys before the trial rollout of eSyM to inform development and implementation. Stakeholders included:
  * patient advisory councils
  * health system leaders
  * clinicians
  * clinic support staff/administration
  * IT/Informatics
  Interventions: Other: Stakeholder Survey (Control Period)
- Stakeholder Feedback (Intervention Period) (Other): Eligible stakeholders at each SIMPRO site were invited to provide feedback through surveys after the trial rollout of eSyM to inform intervention normalization and sustainability. Stakeholders included:
  * health system leaders
  * clinicians
  * clinic support staff/administration
  * IT/Informatics
  Interventions: Other: Stakeholder Survey (Intervention Period)
- SASS Questionnaire Participants (Control Period) (Other): A subset of trial control patients were asked to complete a research questionnaire called the SASS Questionnaire before the roll-out of eSyM to assess patient outcomes including self-efficacy, attainment of informational needs, symptom burden, and satisfaction with care.
  Interventions: Other: SASS Questionnaire
- SASS Questionnaire Participants (Intervention Period) (Other): A subset of trial intervention patients were asked to complete a research questionnaire called the SASS Questionnaire after the roll-out of eSyM to assess patient outcomes including self-efficacy, attainment of informational needs, symptom burden, and satisfaction with care.
  Interventions: Other: SASS Questionnaire
- Patient Qualitative Interviews (Other): A subset of trial intervention patients were asked to participate in a one-time patient interview to provide feedback on facilitators and barriers to eSyM implementation and adoption after the roll-out of eSyM.
  Interventions: Other: Qualitative Interview
- Stakeholder Qualitative Interviews (Other): A subset of eligible stakeholders at each site were asked to participate in a one-time interview to provide feedback on facilitators and barriers to eSyM implementation and adoption after the roll-out of eSyM.
  Interventions: Other: Qualitative Interview
- Pilot Testing (Other): A subset of control patients at each site were selected to pilot test the eSyM intervention prior to trial start.
  Interventions: Other: eSyM
- Cluster Randomized Trial (Control Patients) (No Intervention): These patients (and/or proxy) were seen at a participating site prior to the trial rollout of eSyM and were not exposed to the eSyM intervention.
- Cluster Randomized Trial (Intervention Patients) (Experimental): These patients (and/or proxy) were seen at a participating site after the trial rollout of eSyM and were exposed to the eSyM intervention.
  Interventions: Other: eSyM

INTERVENTIONS:
Other: Stakeholder Survey (Control Period) — Before eSyM go-live, study team members from each site will solicit input via emailed survey, remote meetings and/or in-person meeting on the use of ePROs in oncology from stakeholders to obtain input regarding adaptation, anticipated challenges, and implementation.
  Arms: Stakeholder Feedback (Control Period)
Other: Stakeholder Survey (Intervention Period) — After eSyM go-live and on an ongoing basis, we will evaluate the implementation process at each of the sites with a focus on adoption, appropriateness, acceptability, sustainability, penetration, and scalability. We will do so through emailed surveys and/or discussions with health system leadership, clinicians, clinic support staff, and informatics/IT staff.
  Arms: Stakeholder Feedback (Intervention Period)
Other: Qualitative Interview — A small subset of patients and stakeholders were invited to take part in qualitative interviews after the eSyM trial rollout.
  Arms: Patient Qualitative Interviews; Stakeholder Qualitative Interviews
Other: SASS Questionnaire — A subset of control and intervention patients will be asked to complete a research questionnaire called the "SASS Questionnaire" asking about their Self-efficacy, Attainment of information needs, Symptom burden, and Satisfaction with care.
  Arms: SASS Questionnaire Participants (Control Period); SASS Questionnaire Participants (Intervention Period)
Other: eSyM — The electronic symptom management (eSyM) program is the EHR-integrated ePRO program being evaluated through this trial.
  Arms: Cluster Randomized Trial (Intervention Patients); Pilot Testing

SUMMARY:
Deficits in the management of common symptoms cause substantial morbidity for cancer patients.Because the health care delivery system is structured to be reactive and not proactive, there are missed opportunities to optimize symptom control. Growth in Internet access and proliferation of smartphones has created an opportunity to re-engineer cancer care delivery. Electronic symptom tracking and feedback is a promising strategy to improve symptom control. Electronic patient reported outcome (ePRO) monitoring of cancer symptoms has been shown to decrease symptom burden, improve quality of life, reduce acute care and even extend survival. SIMPRO will use functioning ePRO prototypes to create and refine the electronic symptom management system eSyM

DETAILED DESCRIPTION:
A multi-disciplinary team of investigators from 6 health systems have formed the Symptom Management IMplementation of Patient Reported Outcomes in Oncology (SIMPRO) Research Center. SIMPRO will use functioning ePRO prototypes to create and refine the electronic symptom management system eSyM. eSyM is the name of the platform the team will refine, integrate, implement and evaluate. eSyM addresses each of the 4 evidence gaps by:

* Implementing eSyM in cancer centers in small, rural or community-based systems.
* Integrating eSyM into the EHR (electronic health record) of the predominant vendor used nationwide.
* Leveraging evidence-based tools, patient engagement, and population management.
* Executing this work using the Consolidated Framework for Implementation Research across all phases to maximize the chances that eSyM and similar systems achieve their intended goals and decrease the morbidity of cancer treatment at a population level.

This project contains 5 activities:

1. Obtain stakeholder feedback
2. Build and deploy eSyM
3. Pilot test eSyM
4. Pragmatic stepped-wedge cluster randomized trial
5. Integration of eSyM data to develop algorithms to estimate the risk of experiencing an outcome, including, but not limited to, ED usage and hospitalization among cancer patients

ELIGIBILITY:
Inclusion Criteria:

Stakeholder Feedback and Stakeholder Qualitative Interviews Population:

* Age ≥ 18 years
* The potential stakeholders are: patient advisory council members, health system leaders, clinicians, clinic support staff/administration, IT/Informatics staff

Cluster Randomized Trial, Patient QualitativeInterviews, Pilot Testing & SASS Questionnaire Population:

* Age ≥ 18 years
* Priority population will be patients who meet one of the following:

  * Suspected thoracic cancer [lung or bronchus] AND is inpatient following thoracic surgery.
  * Suspected gastrointestinal cancer [colorectal, pancreas, liver/biliary, esophagus,or gastric] AND is inpatient following gastrointestinal surgery.
  * Suspected gynecologic cancer [ovary, uterus, or cervix] AND is inpatient following gynecologic surgery.
  * Diagnosis of thoracic cancer [lung or bronchus] AND scheduled to start a new treatment plan for thoracic cancer.
  * Diagnosis of gastrointestinal cancer [colorectal, pancreas, liver/biliary, esophagus,or gastric] AND scheduled to start a new treatment plan for gastrointestinal cancer.
  * Diagnosis of gynecologic cancer [ovary, uterus, or cervix] AND scheduled to start a new treatment plan for gynecologic cancer.
* Total population allowed to use eSyM:

  * Any patient at any participating site.

Exclusion Criteria:

- Participants not meeting the inclusion critera above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42808 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2025-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hassett, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (6):
- United States (6):
  - Maine Medical Center, Portland, Maine
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Brown University Health (formerly Lifespan Cancer Institute), Providence, Rhode Island
  - Baptist Memoiral HealthCare, Memphis, Tennessee
  - West Virginia University Medical Center, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research data set used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: DFCI (Dana-Farber Cancer Institute) - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer Statistics, 2017. CA Cancer J Clin. 2017 Jan;67(1):7-30. doi: 10.3322/caac.21387. Epub 2017 Jan 5. PMID 28055103
- [Background] Cleeland CS. Symptom burden: multiple symptoms and their impact as patient-reported outcomes. J Natl Cancer Inst Monogr. 2007;(37):16-21. doi: 10.1093/jncimonographs/lgm005. PMID 17951226
- [Background] Hofman M, Ryan JL, Figueroa-Moseley CD, Jean-Pierre P, Morrow GR. Cancer-related fatigue: the scale of the problem. Oncologist. 2007;12 Suppl 1:4-10. doi: 10.1634/theoncologist.12-S1-4. PMID 17573451
- [Background] Teunissen SC, Wesker W, Kruitwagen C, de Haes HC, Voest EE, de Graeff A. Symptom prevalence in patients with incurable cancer: a systematic review. J Pain Symptom Manage. 2007 Jul;34(1):94-104. doi: 10.1016/j.jpainsymman.2006.10.015. Epub 2007 May 23. PMID 17509812
- [Background] Temel JS, Pirl WF, Lynch TJ. Comprehensive symptom management in patients with advanced-stage non-small-cell lung cancer. Clin Lung Cancer. 2006 Jan;7(4):241-9. doi: 10.3816/CLC.2006.n.001. PMID 16512977
- [Background] Janjan N. Palliation and supportive care in radiation medicine. Hematol Oncol Clin North Am. 2006 Feb;20(1):187-211. doi: 10.1016/j.hoc.2006.01.010. PMID 16580563
- [Background] Fleishman SB. Treatment of symptom clusters: pain, depression, and fatigue. J Natl Cancer Inst Monogr. 2004;(32):119-23. doi: 10.1093/jncimonographs/lgh028. PMID 15263052
- [Background] Hernandez-Boussard T, Graham LA, Desai K, Wahl TS, Aucoin E, Richman JS, Morris MS, Itani KM, Telford GL, Hawn MT. The Fifth Vital Sign: Postoperative Pain Predicts 30-day Readmissions and Subsequent Emergency Department Visits. Ann Surg. 2017 Sep;266(3):516-524. doi: 10.1097/SLA.0000000000002372. PMID 28657940
- [Background] Kenzik KM, Ganz PA, Martin MY, Petersen L, Hays RD, Arora N, Pisu M. How much do cancer-related symptoms contribute to health-related quality of life in lung and colorectal cancer patients? A report from the Cancer Care Outcomes Research and Surveillance (CanCORS) Consortium. Cancer. 2015 Aug 15;121(16):2831-9. doi: 10.1002/cncr.29415. Epub 2015 Apr 17. PMID 25891437
- [Background] Hassett MJ, Wong S, Osarogiagbon RU, Bian J, Dizon DS, Jenkins HH, Uno H, Cronin C, Schrag D; SIMPRO Co-Investigators. Implementation of patient-reported outcomes for symptom management in oncology practice through the SIMPRO research consortium: a protocol for a pragmatic type II hybrid effectiveness-implementation multi-center cluster-randomized stepped wedge trial. Trials. 2022 Jun 16;23(1):506. doi: 10.1186/s13063-022-06435-1. PMID 35710449
- [Result] Hassett MJ, Cronin C, Tsou TC, Wedge J, Bian J, Dizon DS, Hazard-Jenkins H, Osarogiagbon RU, Wong S, Basch E, Austin T, McCleary N, Schrag D. eSyM: An Electronic Health Record-Integrated Patient-Reported Outcomes-Based Cancer Symptom Management Program Used by Six Diverse Health Systems. JCO Clin Cancer Inform. 2022 Jan;6:e2100137. doi: 10.1200/CCI.21.00137. PMID 34985914
- [Result] Paudel R, Enzinger AC, Uno H, Cronin C, Wong SL, Dizon DS, Hazard Jenkins H, Bian J, Osarogiagbon RU, Jensen RE, Mitchell SA, Schrag D, Hassett MJ. Effects of a change in recall period on reporting severe symptoms: an analysis of a pragmatic multisite trial. J Natl Cancer Inst. 2024 Jul 1;116(7):1137-1144. doi: 10.1093/jnci/djae049. PMID 38445744
- [Result] Paudel R, Tramontano AC, Cronin C, Wong SL, Dizon DS, Jenkins HH, Bian J, Osarogiagbon RU, Schrag D, Hassett MJ. Assessing Patient Readiness for an Electronic Patient-Reported Outcome-Based Symptom Management Intervention in a Multisite Study. JCO Oncol Pract. 2024 Jan;20(1):77-84. doi: 10.1200/OP.23.00339. Epub 2023 Nov 27. PMID 38011613
- [Result] Ivatury SJ, Hazard-Jenkins HW, Brooks GA, McCleary NJ, Wong SL, Schrag D. Translation of Patient-Reported Outcomes in Oncology Clinical Trials to Everyday Practice. Ann Surg Oncol. 2020 Jan;27(1):65-72. doi: 10.1245/s10434-019-07749-2. Epub 2019 Aug 26. PMID 31452053
- [Result] Phillips JD, Wong SL. Patient-Reported Outcomes in Surgical Oncology: An Overview of Instruments and Scores. Ann Surg Oncol. 2020 Jan;27(1):45-53. doi: 10.1245/s10434-019-07752-7. Epub 2019 Aug 28. PMID 31463699
- [Result] Hassett M, Dias S, Cronin C, Schrag D, McCleary N, Simpson J, Poirier-Shelton T, Bian J, Reich J, Dizon D, Begnoche M, Jenkins HH, Tasker L, Wong S, Pearson L, Paudel R, Osarogiagbon RU. Strategies for implementing an electronic patient-reported outcomes-based symptom management program across six cancer centers. BMC Health Serv Res. 2024 Nov 12;24(1):1386. doi: 10.1186/s12913-024-11536-5. PMID 39533260
- [Result] Paudel R, Dias S, Wade CG, Cronin C, Hassett MJ. Use of Patient-Reported Outcomes in Risk Prediction Model Development to Support Cancer Care Delivery: A Scoping Review. JCO Clin Cancer Inform. 2024 Nov;8:e2400145. doi: 10.1200/CCI-24-00145. Epub 2024 Nov 1. PMID 39486014
- [Result] Mallow J, Bailey A, Tasker L, Hazard H, Hassett M, Cronin C, Paudel R, Bian J, Dizon DS, Osarogiagbon RU, Schrag D, Wong SL. Perceptions of an Electronic Patient Symptom Reporting Tool by Clinicians. Comput Inform Nurs. 2026 Jan 1;44(1):e01313. doi: 10.1097/CIN.0000000000001313. PMID 40257368
- [Result] Beqari J, Hurd J, Tramontano AC, Cronin C, Potter A, Wong S, Schrag D, Dizon DS, Bian J, Osarogiagbon RU, Hazard-Jenkins H, Phillips JD, Abbas AE, Warikoo IM, Anderson M, Seastedt KP, Lanuti M, Colson YL, Wright CD, Hassett M, Jeffrey Yang CF. The implementation of an electronic symptom management system to monitor postoperative pain in thoracic surgery patients: A multicenter evaluation. JTCVS Open. 2025 Feb 25;25:485-499. doi: 10.1016/j.xjon.2025.02.010. eCollection 2025 Jun. PMID 40631021
- [Result] Cronin, C., Barrett, F., Dias, S., Wong, S. L., Pearson, L., Hazard-Jenkins, H., Bian, J. J., Dizon, D. S., Osarogiagbon, R. U., Schrag, D., & Hassett, M. J. (2024). Electronic Patient-Reported Outcomes in Oncology: Lessons from Six Cancer Centers. NEJM Catalyst Innovations in Care Delivery, 5(2). https://doi.org/10.1056/cat.23.0331
- [Derived] Kuharic M, Merle JL, Cella D, Mitchell SA, DiMartino L, Ridgeway JL, Dizon DS, Paudel R, Austin JD, Wong SL, Flores AM, Cheville AL, Smith JD; IMPACT Consortium. Psychometric evaluation of the NoMAD instrument in cancer care settings: assessing factorial validity, measurement invariance, and differential item functioning. Implement Sci Commun. 2025 Jun 16;6(1):72. doi: 10.1186/s43058-025-00756-3. PMID 40524282

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients and stakeholders were recruited at the six participating sites between Jan. 2018 and Feb. 2023. As this was a stepped wedge trial, each period has distinct enrollment.
  For the entire trial, grand total enrollment was 39,942 patients (21,112 control patients and 18,830 intervention patients).
Groups:
- Medical Oncology eSyM Site 1: Periods 1-2: Transition phase with control & intervention participants enrolled Periods 3-7: eSyM Intervention participants enrolled
- Surgical eSyM Site 1: Period 1-6: No eSyM Intervention (Control Period) Period 7: Transition phase with control and intervention participants enrolled
- Medical Oncology eSyM Site 2: Periods 1-2: No eSyM Intervention (Control Period) Period 3: Transition phase with both control and intervention participants enrolled Periods 4-7: eSyM Intervention Period
- Surgical eSyM Site 2: Periods 1-5: No eSyM Intervention (Control Period) Periods 6: Transition phase with both control and intervention participants enrolled Period 7: eSyM intervention participants enrolled
- Medical Oncology eSyM Site 3: Periods 1-3: No eSyM Intervention (Control Period) Period 4: Transition phase with both control and intervention participants enrolled Periods 5-7: eSyM Intervention Period
- Surgical eSyM Site 3: Periods 1-4: No eSyM Intervention (Control Period) Period 5: Transition phase with control and intervention participants enrolled Periods 6-7: eSyM Intervention Period
- Medical Oncology eSyM Site 4: Periods 1-5: No eSyM Intervention (Control Period) Period 6: Transition phase with control and intervention participants enrolled Periods 7: eSyM Intervention Period
- Surgical eSyM Site 4: Periods 1-3: No eSyM Intervention (Control Period) Period 4: Transition phase with control and intervention participants enrolled Periods 5-7: eSyM Intervention Period
- Medical Oncology eSyM Site 5: Periods 1-5: No eSyM Intervention (Control Period) Period 6: Transition phase with control and intervention participants enrolled Period 7: eSyM Intervention Period
- Surgical eSyM Site 5: Periods 1-2: No eSyM Intervention (Control Period) Period 3: Transition phase with control and intervention participants enrolled Periods 4-7: eSyM Intervention Period
- Medical Oncology eSyM Site 6: Periods 1-6: No eSyM Intervention (Control Period) Periods 7: Transition phase with control and intervention participants
- Surgical eSyM Site 6: Periods 1: No eSyM Intervention (Control Period) Period 2: Transition phase with control and intervention participants enrolled Periods 3-7: eSyM Intervention Period
Period: Period 1 (June 2018-August 2019)
Arm/Group | Medical Oncology eSyM Site 1 | Surgical eSyM Site 1 | Medical Oncology eSyM Site 2 | Surgical eSyM Site 2 | Medical Oncology eSyM Site 3 | Surgical eSyM Site 3 | Medical Oncology eSyM Site 4 | Surgical eSyM Site 4 | Medical Oncology eSyM Site 5 | Surgical eSyM Site 5 | Medical Oncology eSyM Site 6 | Surgical eSyM Site 6
Started | 1078 (During this transition phase, there were 1075 control and 3 intervention participants (total = 1078 participants).) | 957 | 321 | 954 | 881 | 3219 | 105 | 690 | 134 | 549 | 303 | 1065
Completed | 1078 (During this transition phase, there were 1075 control and 3 intervention participants (total = 1078 participants).) | 957 | 321 | 954 | 881 | 3219 | 105 | 690 | 134 | 549 | 303 | 1065
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2 (September 2019-February 2020)
Arm/Group | Medical Oncology eSyM Site 1 | Surgical eSyM Site 1 | Medical Oncology eSyM Site 2 | Surgical eSyM Site 2 | Medical Oncology eSyM Site 3 | Surgical eSyM Site 3 | Medical Oncology eSyM Site 4 | Surgical eSyM Site 4 | Medical Oncology eSyM Site 5 | Surgical eSyM Site 5 | Medical Oncology eSyM Site 6 | Surgical eSyM Site 6
Started | 608 (During this transition phase, there were 18 control and 590 intervention participants (total = 608 participants).) | 286 | 213 | 360 | 305 | 1537 | 78 | 288 | 54 | 478 | 100 | 496 (During this transition phase, there were 166 control and 330 intervention participants (total = 496 participants))
Completed | 608 (During this transition phase, there were 18 control and 590 intervention participants (total = 608 participants)) | 286 | 213 | 360 | 305 | 1537 | 78 | 288 | 54 | 478 | 100 | 496 (During this transition phase, there were 166 control and 330 intervention participants (total = 496 participants))
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3 (March 2020-August 2020)
Arm/Group | Medical Oncology eSyM Site 1 | Surgical eSyM Site 1 | Medical Oncology eSyM Site 2 | Surgical eSyM Site 2 | Medical Oncology eSyM Site 3 | Surgical eSyM Site 3 | Medical Oncology eSyM Site 4 | Surgical eSyM Site 4 | Medical Oncology eSyM Site 5 | Surgical eSyM Site 5 | Medical Oncology eSyM Site 6 | Surgical eSyM Site 6
Started | 434 | 310 | 205 (During this transition phase, there were 11 control and 194 intervention participants (total = 205 participants)) | 52 | 336 | 1138 | 65 | 257 | 59 | 516 (During this transition phase, there were 143 control and 373 intervention participants (total = 516 participants)) | 64 | 430
Completed | 434 | 310 | 205 (During this transition phase, there were 11 control and 194 intervention participants (total = 205 participants)) | 52 | 336 | 1138 | 65 | 257 | 59 | 516 (During this transition phase, there were 143 control and 373 intervention participants (total = 516 participants)) | 64 | 430
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 4 (September 2020-February 2021)
Arm/Group | Medical Oncology eSyM Site 1 | Surgical eSyM Site 1 | Medical Oncology eSyM Site 2 | Surgical eSyM Site 2 | Medical Oncology eSyM Site 3 | Surgical eSyM Site 3 | Medical Oncology eSyM Site 4 | Surgical eSyM Site 4 | Medical Oncology eSyM Site 5 | Surgical eSyM Site 5 | Medical Oncology eSyM Site 6 | Surgical eSyM Site 6
Started | 380 | 310 | 196 | 14 | 339 (During this transition phase, there were 39 control and 300 intervention participants (total = 339 participants)) | 1404 | 94 | 375 (During this transition phase, there were 257 control and 118 intervention participants (total = 375 participants)) | 62 | 545 | 95 | 419
Completed | 380 | 310 | 196 | 14 | 339 (During this transition phase, there were 39 control and 300 intervention participants (total = 339 participants)) | 1404 | 94 | 375 (During this transition phase, there were 257 control and 118 intervention participants (total = 375 participants)) | 62 | 545 | 95 | 419
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 5 (March 2021-August 2021)
Arm/Group | Medical Oncology eSyM Site 1 | Surgical eSyM Site 1 | Medical Oncology eSyM Site 2 | Surgical eSyM Site 2 | Medical Oncology eSyM Site 3 | Surgical eSyM Site 3 | Medical Oncology eSyM Site 4 | Surgical eSyM Site 4 | Medical Oncology eSyM Site 5 | Surgical eSyM Site 5 | Medical Oncology eSyM Site 6 | Surgical eSyM Site 6
Started | 433 | 323 | 177 | 79 | 349 | 961 (During this transition phase, there were 496 control and 465 intervention participants (total = 961 participants)) | 261 | 254 | 126 | 534 | 106 | 485
Completed | 433 | 323 | 177 | 79 | 349 | 961 (During this transition phase, there were 496 control and 465 intervention participants (total = 961 participants)) | 261 | 254 | 126 | 534 | 106 | 485
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 6 (September 2021-February 2022)
Arm/Group | Medical Oncology eSyM Site 1 | Surgical eSyM Site 1 | Medical Oncology eSyM Site 2 | Surgical eSyM Site 2 | Medical Oncology eSyM Site 3 | Surgical eSyM Site 3 | Medical Oncology eSyM Site 4 | Surgical eSyM Site 4 | Medical Oncology eSyM Site 5 | Surgical eSyM Site 5 | Medical Oncology eSyM Site 6 | Surgical eSyM Site 6
Started | 359 | 382 | 121 | 339 (During this transition phase, there were 150 control and 189 intervention participants (total = 339 participants)) | 332 | 991 | 299 (During this transition phase, there were 22 control and 277 intervention participants (total = 299 participants)) | 286 | 144 (During this transition phase, there were 83 control and 61 intervention participants (total = 144 participants)) | 395 | 115 | 436
Completed | 359 | 382 | 121 | 339 (During this transition phase, there were 150 control and 189 intervention participants (total = 339 participants)) | 332 | 991 | 299 (During this transition phase, there were 22 control and 277 intervention participants (total = 299 participants)) | 286 | 144 (During this transition phase, there were 83 control and 61 intervention participants (total = 144 participants)) | 395 | 115 | 436
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 7 (March 2022-February 2023)
Arm/Group | Medical Oncology eSyM Site 1 | Surgical eSyM Site 1 | Medical Oncology eSyM Site 2 | Surgical eSyM Site 2 | Medical Oncology eSyM Site 3 | Surgical eSyM Site 3 | Medical Oncology eSyM Site 4 | Surgical eSyM Site 4 | Medical Oncology eSyM Site 5 | Surgical eSyM Site 5 | Medical Oncology eSyM Site 6 | Surgical eSyM Site 6
Started | 697 | 662 (During this transition phase, there were 98 control and 564 intervention participants (total = 662 participants)) | 276 | 654 | 768 | 2000 | 544 | 689 | 334 | 680 | 230 (During this transition phase, there were 25 control and 205 intervention participants (total = 230 participants)) | 963
Completed | 697 | 662 (During this transition phase, there were 98 control and 564 intervention participants (total = 662 participants)) | 276 | 654 | 768 | 2000 | 544 | 689 | 334 | 680 | 230 (During this transition phase, there were 25 control and 205 intervention participants (total = 230 participants)) | 963
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Please note: demographics for both medical oncology and surgical patients are combined because the primary analysis evaluated the entire cohort combined together. The pre-specified analysis plan in the study protocol was to report baseline characteristics data for medical oncology and surgery combined.
Groups:
- eSyM Control Participants (Medical Oncology and Surgery Participants Combined): These patients (and/or proxy) were seen at a participating site prior to the trial rollout of eSyM and were not exposed to the eSyM intervention.
  This group includes the following trial subsets:
  * patients NOT exposed to the eSyM intervention through the stepped wedge cluster randomized trial (control cohort)
  * patients participating in the SASS control questionnaire
  Please note: demographics for both medical oncology and surgical patients are combined because the primary analysis evaluated the entire cohort combined together.
- eSyM Intervention Participants (Medical Oncology and Surgery Participants Combined): These patients (and/or proxy) were seen at a participating site after the trial rollout of eSyM and were exposed to the eSyM intervention.
  This group includes the following trial subsets:
  * patients exposed to the eSyM intervention through the stepped wedge cluster randomized trial (intervention cohort)
  * patients participating in the SASS intervention questionnaire
  * patients participating in qualitative interviews
  * patients participating in pilot testing
  Please note: demographics for both medical oncology and surgical patients are combined because the primary analysis evaluated the entire cohort combined together.
- Total: Total of all reporting groups
Arm/Group | eSyM Control Participants (Medical Oncology and Surgery Participants Combined) | eSyM Intervention Participants (Medical Oncology and Surgery Participants Combined) | Total
Number analyzed (Participants) | 21,112 | 18,830 | 39942
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 62 [51 to 71] | 65 [55 to 72] | 63 [53 to 72]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 14273 | 11929 | 26202
  Male | 6837 | 6900 | 13737
  Other | 2 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 808 | 516 | 1324
  Non-Hispanic Black | 2024 | 1378 | 3402
  Non-Hispanic White | 16903 | 15848 | 32751
  Other | 1377 | 1088 | 2465

OUTCOME MEASURES:

1. Primary Outcome: Emergency Department Treat/Release [EDTR] Event Occurrence Status at Day 30
Description: The primary study outcome of the stepped wedge cluster RCT (randomized controlled trial) is the EDTR rate. This outcome will be defined in relation to the date of discharge from hospital (surgical cohort) or the initiation date of a new intravenous chemo regimen (medical oncology cohort). This is a binary outcome and we will analyze the absolute difference and odds ratio for the medical oncology and surgical cohorts combined and independently.
Time Frame: 30 days
Population: The primary analysis included data from both medical oncology and surgery. As a secondary analysis, we analyzed the data from MO and Surg separately and estimated the intervention effect for each outcome. Results for both combined and separate analyses are reported below.
Measure: Number; unit: percentage of patients with event
Arm/Group | Cluster Randomized Trial (Control Patients) | Cluster Randomized Trial (Intervention Patients)
Number analyzed (Participants) | 21112 | 18830
percentage of patients with event
  Medical Oncology Cohort: number analyzed (Participants) | 5150 | 7030
  Medical Oncology Cohort | 5.8 | 6.9
  Surgery Cohort: number analyzed (Participants) | 15962 | 11800
  Surgery Cohort | 5.3 | 5.8
  Medical Oncology + Surgery Combined Cohort | 5.4 | 6.2
Statistical Analysis 1: Comparison: Cluster Randomized Trial (Control Patients) vs Cluster Randomized Trial (Intervention Patients); Adjusted analysis comparing control versus intervention patients (chemo and surgical patients combined); Test type: Superiority; p = 0.214, Regression, Logistic; Odds Ratio (OR) = 1.104, 95% CI 2-sided [0.944 to 1.290]
Statistical Analysis 2: Comparison: Cluster Randomized Trial (Control Patients) vs Cluster Randomized Trial (Intervention Patients); Adjusted analysis comparing control versus intervention patients (medical oncology patients only); Test type: Superiority; p = 0.565, Regression, Logistic; Odds Ratio (OR) = 0.927, 95% CI 2-sided [0.715 to 1.201]
Statistical Analysis 3: Comparison: Cluster Randomized Trial (Control Patients) vs Cluster Randomized Trial (Intervention Patients); Adjusted analysis comparing control versus intervention patients (surgical patients only); Test type: Superiority; p = 0.042, Regression, Logistic; Odds Ratio (OR) = 1.225, 95% CI 2-sided [1.008 to 1.490]

2. Secondary Outcome: Emergency Department Treat/Release [EDTR] Event Occurrence Status at Day 90
Description: This outcome will be defined in relation to the date of discharge from hospital (surgical cohort) or the initiation date of a new intravenous chemo regimen (medical oncology cohort). This is a binary outcome and we will analyze the absolute difference and odds ratio for the medical oncology and surgical cohorts combined and independently.
Time Frame: 90 days
Population: as for outcome 1
Measure: Number; unit: percentage of patients with event
Arm/Group | Cluster Randomized Trial (Control Patients) | Cluster Randomized Trial (Intervention Patients)
Number analyzed (Participants) | 21112 | 18830
percentage of patients with event
  Medical Oncology: number analyzed (Participants) | 5150 | 7030
  Medical Oncology | 11.6 | 13.8
  Surgery: number analyzed (Participants) | 15962 | 11800
  Surgery | 8.8 | 9.7
  Medical Oncology + Surgery | 9.5 | 11.2
Statistical Analysis 1: Comparison: Cluster Randomized Trial (Control Patients) vs Cluster Randomized Trial (Intervention Patients); Adjusted analysis comparing control versus intervention patients (medical oncology and surgical patients combined); Test type: Other; p = 0.050, Regression, Logistic; Odds Ratio (OR) = 1.128, 95% CI 2-sided [1.000 to 1.272]
Statistical Analysis 2: Comparison: Cluster Randomized Trial (Control Patients) vs Cluster Randomized Trial (Intervention Patients); Adjusted analysis comparing control versus intervention patients (medical oncology patients only); Test type: Other; p = 0.903, Regression, Logistic; Odds Ratio (OR) = 1.012, 95% CI 2-sided [0.836 to 1.225]
Statistical Analysis 3: Comparison: Cluster Randomized Trial (Control Patients) vs Cluster Randomized Trial (Intervention Patients); Adjusted analysis comparing control versus intervention patients (surgical patients only); Test type: Other; p = 0.014, Regression, Logistic; Odds Ratio (OR) = 1.215, 95% CI 2-sided [1.040 to 1.418]

3. Secondary Outcome: Admissions Event Occurrence Status at Day 30
Description: as for outcome 2
Time Frame: 30 Days
Population: as for outcome 1
Measure: Number; unit: percentage of patients with event
Groups:
- Cluster Randomized Trial (Control Patients): These patients (and/or proxy) were seen at a participating site prior to the trial rollout of eSyM and were not exposed to the eSyM intervention.
  This group includes the following trial subsets:
  * patients NOT exposed to the eSyM intervention through the stepped wedge cluster randomized trial (control cohort)
  * patients participating in the SASS control questionnaire
- Cluster Randomized Trial (Intervention Patients): These patients (and/or proxy) were seen at a participating site after the trial rollout of eSyM and were exposed to the eSyM intervention.
  This group includes the following trial subsets:
  * patients exposed to the eSyM intervention through the stepped wedge cluster randomized trial (intervention cohort)
  * patients participating in the SASS intervention questionnaire
  * patients participating in qualitative interviews
  * patients participating in pilot testing
Arm/Group | Cluster Randomized Trial (Control Patients) | Cluster Randomized Trial (Intervention Patients)
Number analyzed (Participants) | 21112 | 18830
percentage of patients with event
  Medical Oncology: number analyzed (Participants) | 5150 | 7030
  Medical Oncology | 10.8 | 10.7
  Surgery: number analyzed (Participants) | 15962 | 11800
  Surgery | 7.7 | 8.2
  Medical Oncology + Surgery | 8.5 | 9.1
Statistical Analysis 1: Comparison: Cluster Randomized Trial (Control Patients) vs Cluster Randomized Trial (Intervention Patients); Adjusted analysis comparing control versus intervention patients (medical oncology and surgical patients combined); Test type: Other; p = 0.978, Regression, Logistic; Odds Ratio (OR) = 1.002, 95% CI 2-sided [0.881 to 1.139]
Statistical Analysis 2: Comparison: Cluster Randomized Trial (Control Patients) vs Cluster Randomized Trial (Intervention Patients); Adjusted analysis comparing control versus intervention patients (medical oncology patients only); Test type: Other; p = 0.126, Regression, Logistic; Odds Ratio (OR) = 0.854, 95% CI 2-sided [0.697 to 1.046]
Statistical Analysis 3: Comparison: Cluster Randomized Trial (Control Patients) vs Cluster Randomized Trial (Intervention Patients); Adjusted analysis comparing control versus intervention patients (surgical patients only); Test type: Other; p = 0.254, Regression, Logistic; Odds Ratio (OR) = 1.102, 95% CI 2-sided [0.933 to 1.302]

4. Secondary Outcome: Admissions Event Occurrence Status at Day 90
Description: as for outcome 2
Time Frame: 90 Days
Population: as for outcome 1
Measure: Number; unit: percentage of patients with event
Arm/Group | Cluster Randomized Trial (Control Patients) | Cluster Randomized Trial (Intervention Patients)
Number analyzed (Participants) | 21112 | 18830
percentage of patients with event
  Medical Oncology: number analyzed (Participants) | 5150 | 7030
  Medical Oncology | 20.8 | 21.9
  Surgery: number analyzed (Participants) | 15962 | 11800
  Surgery | 12.8 | 13.1
  Medical Oncology + Surgery | 14.7 | 16.4
Statistical Analysis 1: Comparison: Cluster Randomized Trial (Control Patients); Adjusted analysis comparing control versus intervention patients (medical oncology and surgical patients combined); Test type: Other; p = 0.209, Regression, Logistic; Odds Ratio (OR) = 1.068, 95% CI 2-sided [0.964 to 1.183]
Statistical Analysis 2: Comparison: Cluster Randomized Trial (Control Patients) vs Cluster Randomized Trial (Intervention Patients); Adjusted analysis comparing control versus intervention patients (medical oncology patients only); Test type: Other; p = 0.924, Regression, Logistic; Odds Ratio (OR) = 0.992, 95% CI 2-sided [0.850 to 1.159]
Statistical Analysis 3: Comparison: Cluster Randomized Trial (Control Patients) vs Cluster Randomized Trial (Intervention Patients); Adjusted analysis comparing control versus intervention patients (surgical patients only); Test type: Other; p = 0.099, Regression, Logistic; Odds Ratio (OR) = 1.122, 95% CI 2-sided [0.979 to 1.286]

5. Secondary Outcome: Difference in Fatigue PROMIS Scores Reported by Participants Before and After eSyM Exposure
Description: Difference in PROMIS fatigue scores between the pre-live and post-live eSyM cohorts. Since the two cohorts were comprised of different patients, comparisons were performed at the population level using mean T-scores. Fatigue was assessed using the PROMIS Fatigue 4-item short form with responses converted to T-scores (score range: 50 indicates the population mean with a standard deviation of 10; decrease in score indicates a positive change). All PROMIS items were scored using the standardized scoring tool kit. The differences in mean T-scores and the corresponding 95% confidence intervals (CI) were calculated for each PROMIS item, comparing the post-live versus pre-live cohort. When comparing group-level change in PROMIS scores, even trivial differences can be statistically significant if the sample size is large enough. The threshold to evaluate within-group change or to make a between-group comparison generally ranges between 2 and 6 T-score points (Terwee et al., 2021).
Time Frame: 30-90 days before and after eSyM go-live
Population: Since only a subset of eSyM patients completed the SASS questionnaire which included PROMIS measures, the analyzed population is smaller than other analytic populations. Distinct surveys were given to medical oncology and surgical patients to account for differences in their care, so the analytic cohorts below are distinct. Results for both the medical oncology and surgical subsets are included below.
Measure: Geometric Mean (Standard Deviation); unit: T-Score
Groups:
- SASS Questionnaire Participants (Intervention Period): A subset of trial intervention patients were asked to complete a research questionnaire called the SASS Questionnaire after the roll-out of eSyM to assess the impact on patient outcomes including self-efficacy, attainment of informational needs, symptom burden, and satisfaction with care.
Arm/Group | SASS Questionnaire Participants (Control Period) | SASS Questionnaire Participants (Intervention Period)
Number analyzed (Participants) | 1043 | 1046
T-Score
  Medical Oncology: number analyzed (Participants) | 490 | 535
  Medical Oncology | 57.4 (10.5) | 55.6 (9.8)
  Surgery: number analyzed (Participants) | 553 | 511
  Surgery | 51.1 (10.9) | 49.0 (11.2)
Statistical Analysis 1: Comparison: SASS Questionnaire Participants (Control Period) vs SASS Questionnaire Participants (Intervention Period); Multivariable regression analyses (medical oncology cohort only); Test type: Superiority; p = 0.04, Regression, Linear; Difference = -1.328, 95% CI 2-sided [-2.593 to -0.062]
Statistical Analysis 2: Comparison: SASS Questionnaire Participants (Control Period) vs SASS Questionnaire Participants (Intervention Period); Multivariable regression analyses (surgical cohort only); Test type: Other; p = 0.004, Regression, Logistic; Difference = -1.958, 95% CI 2-sided [-3.269 to -0.646]

6. Secondary Outcome: Difference in Depression PROMIS Scores Reported by Participants Before and After eSyM Exposure
Description: Difference in PROMIS depression scores between the pre-live and post-live eSyM cohorts. Since the two cohorts were comprised of different patients, comparisons were performed at the population level using mean T-scores. Depression was assessed using the PROMIS Emotional Distress-Depression 4-item short form with responses converted to T-scores (score range: 50 indicates the population mean with a standard deviation of 10; decrease in score indicates a positive change). All PROMIS items were scored using the standardized scoring tool kit. The differences in mean T-scores and the corresponding 95% confidence intervals (CI) were calculated for each PROMIS item, comparing the post-live versus pre-live cohort. When comparing group-level change in PROMIS scores, even trivial differences can be statistically significant if the sample size is large enough. The threshold to evaluate within-group change or to make a between-group comparison generally ranges between 2 and 6 T-score points.
Time Frame: 30-90 days before and after eSyM go-live
Population: as for outcome 5
Measure: Geometric Mean (Standard Deviation); unit: T-Score
Arm/Group | SASS Questionnaire Participants (Control Period) | SASS Questionnaire Participants (Intervention Period)
Number analyzed (Participants) | 1043 | 1046
T-Score
  Medical Oncology: number analyzed (Participants) | 490 | 535
  Medical Oncology | 50.0 (9.0) | 48.7 (8.2)
  Surgery: number analyzed (Participants) | 553 | 511
  Surgery | 47.9 (8.5) | 46.0 (7.6)
Statistical Analysis 1: Comparison: SASS Questionnaire Participants (Control Period) vs SASS Questionnaire Participants (Intervention Period); Multivariable regression analyses (medical oncology cohort only); Test type: Superiority; p = 0.09, Regression, Linear; Difference = -0.925, 95% CI 2-sided [-1.985 to 0.136]
Statistical Analysis 2: Comparison: SASS Questionnaire Participants (Control Period) vs SASS Questionnaire Participants (Intervention Period); Multivariable regression analyses (surgical cohort only); Test type: Superiority; p = 0.002, Regression, Linear; Difference = -1.516, 95% CI 2-sided [-2.474 to -0.557]

7. Secondary Outcome: Difference in Anxiety PROMIS Scores Reported by Participants Before and After eSyM Exposure
Description: Difference in PROMIS anxiety scores between the pre-live and post-live eSyM cohorts. Since the two cohorts were comprised of different patients, comparisons were performed at the population level using mean T-scores. Anxiety was assessed using the PROMIS Emotional Distress-Anxiety 4-item short form with responses converted to T-scores (score range: 50 indicates the population mean with a standard deviation of 10; decrease in score indicates a positive change). All PROMIS items were scored using the standardized scoring tool kit. The differences in mean T-scores and the corresponding 95% confidence intervals (CI) were calculated for each PROMIS item, comparing the post-live versus pre-live cohort. When comparing group-level change in PROMIS scores, even trivial differences can be statistically significant if the sample size is large enough. The threshold to evaluate within-group change or to make a between-group comparison generally ranges between 2 and 6 T-score points.
Time Frame: 30-90 days before and after eSyM go-live
Population: as for outcome 5
Measure: Geometric Mean (Standard Deviation); unit: T-Score
Arm/Group | SASS Questionnaire Participants (Control Period) | SASS Questionnaire Participants (Intervention Period)
Number analyzed (Participants) | 1043 | 1046
T-Score
  Medical Oncology: number analyzed (Participants) | 490 | 535
  Medical Oncology | 52.4 (9.8) | 50.2 (9.5)
  Surgery: number analyzed (Participants) | 553 | 511
  Surgery | 49.9 (9.3) | 47.4 (8.8)
Statistical Analysis 1: Comparison: SASS Questionnaire Participants (Control Period) vs SASS Questionnaire Participants (Intervention Period); Multivariable regression analyses (medical oncology cohort only); Test type: Superiority; p = 0.17, Regression, Linear; Difference = -1.767, 95% CI 2-sided [-2.532 to 0.433]
Statistical Analysis 2: Comparison: SASS Questionnaire Participants (Control Period) vs SASS Questionnaire Participants (Intervention Period); Multivariable regression analyses (surgical cohort only); Test type: Superiority; p < 0.0001, Regression, Linear; Difference = -2.198, 95% CI 2-sided [-3.259 to -1.137]

8. Secondary Outcome: Difference in Pain Interference PROMIS Scores Reported by Participants Before and After eSyM Exposure
Description: Difference in PROMIS pain interference scores between the pre-live and post-live eSyM cohorts. Since the two cohorts were comprised of different patients, comparisons were performed at the population level using mean T-scores. Pain interference was assessed using the PROMIS Pain Interference 4-item short form with responses converted to T-scores (score range: 50 indicates the population mean with a standard deviation of 10; decrease in score indicates a positive change). All PROMIS items were scored using the standardized scoring tool kit. The differences in mean T-scores and the corresponding 95% confidence intervals (CI) were calculated for each PROMIS item, comparing the post-live versus pre-live cohort. When comparing group-level change in PROMIS scores, even trivial differences can be statistically significant if the sample size is large enough. The threshold to evaluate within-group change or to make a between-group comparison generally ranges between 2 and 6 T-score points.
Time Frame: 30-90 days before and after eSyM go-live
Population: as for outcome 5
Measure: Geometric Mean (Standard Deviation); unit: T-Score
Arm/Group | SASS Questionnaire Participants (Control Period) | SASS Questionnaire Participants (Intervention Period)
Number analyzed (Participants) | 1043 | 1046
T-Score
  Medical Oncology: number analyzed (Participants) | 490 | 535
  Medical Oncology | 54.0 (10.3) | 52.7 (9.7)
  Surgery: number analyzed (Participants) | 553 | 511
  Surgery | 52.7 (9.8) | 51.8 (9.5)
Statistical Analysis 1: Comparison: SASS Questionnaire Participants (Control Period) vs SASS Questionnaire Participants (Intervention Period); Multivariable regression analyses (medical oncology cohort only); Test type: Superiority; p = 0.2, Regression, Linear; Difference = -0.8084, 95% CI 2-sided [-2.048 to 0.431]
Statistical Analysis 2: Comparison: SASS Questionnaire Participants (Control Period) vs SASS Questionnaire Participants (Intervention Period); Multivariable regression analyses (surgical cohort only); Test type: Superiority; p = 0.27, Regression, Linear; Difference = -0.652, 95% CI 2-sided [-1.800 to 0.496]

9. Secondary Outcome: Difference in Self-Efficacy PROMIS Scores Reported by Participants Before and After eSyM Exposure
Description: Difference in PROMIS self-efficacy scores between pre-live and post-live eSyM cohorts. Since the two cohorts were comprised of different patients, comparisons were performed at the population level using mean T-scores. Self-efficacy was assessed using the PROMIS Self-Efficacy for Managing Symptoms 8-item short form with responses converted to T-scores (score range: 50 indicates the population mean with a standard deviation of 10; decrease in score indicates a positive change). All PROMIS items were scored using the standardized scoring tool kit. The differences in mean T-scores and the corresponding 95% confidence intervals were calculated for each PROMIS item, comparing the post-live versus pre-live cohort. When comparing group-level change in PROMIS scores, even trivial differences can be statistically significant if the sample size is large enough. The threshold to evaluate within-group change or to make a between-group comparison generally ranges between 2 and 6 T-score points.
Time Frame: 30-90 days before and after eSyM go-live
Population: as for outcome 5
Measure: Geometric Mean (Standard Deviation); unit: T-Score
Arm/Group | SASS Questionnaire Participants (Control Period) | SASS Questionnaire Participants (Intervention Period)
Number analyzed (Participants) | 1043 | 1046
T-Score
  Medical Oncology: number analyzed (Participants) | 490 | 535
  Medical Oncology | 47.6 (8.4) | 47.3 (7.6)
  Surgery: number analyzed (Participants) | 553 | 511
  Surgery | 50.1 (8.8) | 50.8 (8.0)
Statistical Analysis 1: Comparison: SASS Questionnaire Participants (Control Period) vs SASS Questionnaire Participants (Intervention Period); Multivariable regression analyses (medical oncology cohort only); Test type: Superiority; p = 0.23, Regression, Linear; Difference = -0.617, 95% CI 2-sided [-1.620 to 0.386]
Statistical Analysis 2: Comparison: SASS Questionnaire Participants (Control Period) vs SASS Questionnaire Participants (Intervention Period); Multivariable regression analyses (surgical cohort only); Test type: Superiority; p = 0.39, Regression, Linear; Difference = 0.434, 95% CI 2-sided [-0.563 to 1.431]

10. Secondary Outcome: Difference in Physical Function PROMIS Scores Reported by Participants Before and After eSyM Exposure
Description: Difference in PROMIS physical function scores between the pre-live and post-live eSyM cohorts. Since the two cohorts were comprised of different patients, comparisons were performed at the population level using mean T-scores. Physical function was assessed using the PROMIS Physical Function 4-item short form with responses converted to T-scores (score range: 50 indicates the population mean with a standard deviation of 10; decrease in score indicates a positive change). All PROMIS items were scored using the standardized scoring tool kit. The differences in mean T-scores and the corresponding 95% confidence intervals (CI) were calculated for each PROMIS item, comparing the post-live versus pre-live cohort. When comparing group-level change in PROMIS scores, even trivial differences can be statistically significant if the sample size is large enough. The threshold to evaluate within-group change or to make a between-group comparison generally ranges between 2 and 6 T-score points).
Time Frame: 30-90 days before and after eSyM go-live
Population: as for outcome 5
Measure: Geometric Mean (Standard Deviation); unit: T-Score
Arm/Group | SASS Questionnaire Participants (Control Period) | SASS Questionnaire Participants (Intervention Period)
Number analyzed (Participants) | 1043 | 1046
T-Score
  Medical Oncology: number analyzed (Participants) | 490 | 535
  Medical Oncology | 42.3 (9.5) | 42.3 (9.0)
  Surgery: number analyzed (Participants) | 553 | 511
  Surgery | 47.9 (8.9) | 47.5 (9.4)
Statistical Analysis 1: Comparison: SASS Questionnaire Participants (Control Period) vs SASS Questionnaire Participants (Intervention Period); Multivariable regression analyses (medical oncology cohort only); Test type: Superiority; p = 0.22, Regression, Linear; Difference = -0.7, 95% CI 2-sided [-1.829 to 0.429]
Statistical Analysis 2: Comparison: SASS Questionnaire Participants (Control Period) vs SASS Questionnaire Participants (Intervention Period); Multivariable regression analyses (surgical cohort only); Test type: Superiority; p = 0.28, Regression, Linear; Difference = -0.58, 95% CI 2-sided [-1.632 to 0.472]

11. Secondary Outcome: Emergency Department Treat/Release [EDTR] Event Occurrence Status at Day 30 (Comparing eSyM Intervention Responders Versus Non-Responders)
Description: The secondary study outcome of the stepped wedge cluster RCT (randomized controlled trial) is the difference in the EDTR rate between eSyM responders and non-responders. This outcome will be defined in relation to the date of discharge from hospital (surgical cohort) or the initiation date of a new intravenous chemo regimen (medical oncology cohort). This is a binary outcome and we will analyze the absolute difference and odds ratio for the medical oncology and surgical cohorts combined and independently.
  NOTE: The total number of intervention participants in this analysis is greater than the number of intervention participants included in the primary analyses (outcomes 1-4). For outcomes outcomes 1-4, we used the patient's first event during the entire study period. To conduct this analysis of eSyM responders, we used the patient's first event during the intervention period. Approximately 10% of patients in this analysis were counted as a control event in the prior analyses.
Time Frame: 30 days
Population: The primary analysis included data from both medical oncology and surgery. As a secondary analysis, we analyzed the data from MO and Surg separately and estimated the intervention effect for each outcome. Results for both combined and separate analyses are reported below.
  NOTE: To conduct this analysis of eSyM responders, we used the patient's first event during the intervention period. Approximately 10% of patients in this analysis were counted as a control event in outcomes 1-4.
Measure: Number; unit: percentage of patients with event
Groups:
- Cluster Randomized Trial (Intervention Patients - eSyM Responders): These patients (and/or proxy) were seen at a participating site after the trial rollout of eSyM. These patients were exposed to eSyM and used it to report symptoms.
- Cluster Randomized Trial (Intervention Patients - eSyM Non-Responders): These patients (and/or proxy) were seen at a participating site after the trial rollout of eSyM. These patients were exposed to eSyM and did NOT use it to report symptoms.
Arm/Group | Cluster Randomized Trial (Intervention Patients - eSyM Responders) | Cluster Randomized Trial (Intervention Patients - eSyM Non-Responders)
Number analyzed (Participants) | 10078 | 10055
percentage of patients with event
  Medical Oncology Cohort: number analyzed (Participants) | 3593 | 4352
  Medical Oncology Cohort | 5.7 | 7.7
  Surgery Cohort: number analyzed (Participants) | 6485 | 5703
  Surgery Cohort | 5.1 | 6.7
  Med Onc + Surgery Combined Cohort | 5.3 | 7.1
Statistical Analysis 1: Comparison: Cluster Randomized Trial (Intervention Patients - eSyM Responders) vs Cluster Randomized Trial (Intervention Patients - eSyM Non-Responders); Adjusted analysis comparing intervention responders versus non-responders (chemo and surgical patients combined); Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 0.842, 95% CI 2-sided [0.776 to 0.913]
Statistical Analysis 2: Comparison: Cluster Randomized Trial (Intervention Patients - eSyM Responders) vs Cluster Randomized Trial (Intervention Patients - eSyM Non-Responders); Adjusted analysis comparing intervention responders versus non-responders (medical oncology patients only); Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 0.780, 95% CI 2-sided [0.688 to 0.885]
Statistical Analysis 3: Comparison: Cluster Randomized Trial (Intervention Patients - eSyM Responders) vs Cluster Randomized Trial (Intervention Patients - eSyM Non-Responders); Adjusted analysis comparing intervention responders versus non-responders (surgical patients only); Test type: Superiority; p = 0.032, Regression, Logistic; Odds Ratio (OR) = 0.889, 95% CI 2-sided [0.799 to 0.990]

12. Secondary Outcome: Emergency Department Treat/Release [EDTR] Event Occurrence Status at Day 90 (Comparing eSyM Intervention Responders Versus Non-Responders)
Description: This outcome will be defined in relation to the date of discharge from hospital (surgical cohort) or the initiation date of a new intravenous chemo regimen (medical oncology cohort). This is a binary outcome and we will analyze the absolute difference and odds ratio for the medical oncology and surgical cohorts combined and independently.
  NOTE: The total number of intervention participants in this analysis is greater than the number of intervention participants included in the primary analyses (outcomes 1-4). For outcomes outcomes 1-4, we used the patient's first event during the entire study period. To conduct this analysis of eSyM responders, we used the patient's first event during the intervention period. Approximately 10% of patients in this analysis were counted as a control event in the prior analyses.
Time Frame: 90 days
Population: as for outcome 11
Measure: Number; unit: percentage of patients with event
Groups:
- Cluster Randomized Trial (Intervention Patients - eSyM Responders): These patients (and/or proxy) were seen at a participating site after trial rollout of eSyM. These patients were exposed to eSyM and used it to report symptoms.
- Cluster Randomized Trial (Intervention Patients - eSyM Non-Responders): These patients (and/or proxy) were seen at a participating site after trial rollout of eSyM. These patients were exposed to eSyM and did not use it to report symptoms.
Arm/Group | Cluster Randomized Trial (Intervention Patients - eSyM Responders) | Cluster Randomized Trial (Intervention Patients - eSyM Non-Responders)
Number analyzed (Participants) | 10078 | 10055
percentage of patients with event
  Medical Oncology: number analyzed (Participants) | 3593 | 4352
  Medical Oncology | 12.1 | 15.1
  Surgery: number analyzed (Participants) | 6485 | 5703
  Surgery | 8.6 | 11.2
  Medical Oncology + Surgery | 9.9 | 12.9
Statistical Analysis 1: Comparison: Cluster Randomized Trial (Intervention Patients - eSyM Responders) vs Cluster Randomized Trial (Intervention Patients - eSyM Non-Responders); Adjusted analysis comparing intervention responders versus non-responders (medical oncology and surgical patients combined); Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 0.893, 95% CI 2-sided [0.839 to 0.949]
Statistical Analysis 2: Comparison: Cluster Randomized Trial (Intervention Patients - eSyM Responders) vs Cluster Randomized Trial (Intervention Patients - eSyM Non-Responders); Adjusted analysis comparing intervention responders versus non-responders (medical oncology patients only); Test type: Superiority; p = 0.003, Regression, Logistic; Odds Ratio (OR) = 0.872, 95% CI 2-sided [0.796 to 0.954]
Statistical Analysis 3: Comparison: Cluster Randomized Trial (Intervention Patients - eSyM Responders) vs Cluster Randomized Trial (Intervention Patients - eSyM Non-Responders); Adjusted analysis comparing intervention responders versus non-responders (surgical patients only); Test type: Superiority; p = 0.027, Regression, Logistic; Odds Ratio (OR) = 0.909, 95% CI 2-sided [0.835 to 0.989]

13. Secondary Outcome: Admissions Event Occurrence Status at Day 30 (Comparing eSyM Intervention Responders Versus Non-Responders)
Description: as for outcome 12
Time Frame: 30 Days
Population: as for outcome 11
Measure: Number; unit: percentage of patients with event
Arm/Group | Cluster Randomized Trial (Intervention Patients - eSyM Responders) | Cluster Randomized Trial (Intervention Patients - eSyM Non-Responders)
Number analyzed (Participants) | 10078 | 10055
percentage of patients with event
  Medical Oncology: number analyzed (Participants) | 3593 | 4352
  Medical Oncology | 7.5 | 12.9
  Surgery: number analyzed (Participants) | 6485 | 5703
  Surgery | 6.2 | 10.5
  Medical Oncology + Surgery | 6.7 | 11.5
Statistical Analysis 1: Comparison: Cluster Randomized Trial (Intervention Patients - eSyM Responders) vs Cluster Randomized Trial (Intervention Patients - eSyM Non-Responders); [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 0.636, 95% CI 2-sided [0.593 to 0.682]
Statistical Analysis 2: Comparison: Cluster Randomized Trial (Intervention Patients - eSyM Responders) vs Cluster Randomized Trial (Intervention Patients - eSyM Non-Responders); Adjusted analysis comparing intervention responders versus non-responders (medical oncology patients only); Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 0.611, 95% CI 2-sided [0.550 to 0.679]
Statistical Analysis 3: Comparison: Cluster Randomized Trial (Intervention Patients - eSyM Responders) vs Cluster Randomized Trial (Intervention Patients - eSyM Non-Responders); Adjusted analysis comparing intervention responders versus non-responders (surgical patients only); Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 0.655, 95% CI 2-sided [0.597 to 0.719]

14. Secondary Outcome: Admissions Event Occurrence Status at Day 90 (Comparing eSyM Intervention Responders Versus Non-Responders)
Description: as for outcome 12
Time Frame: 90 Days
Population: as for outcome 11
Measure: Number; unit: percentage of patients with event
Groups:
- Cluster Randomized Trial (Intervention Patients - eSyM Non-Responders): These patients (and/or proxy) were seen at a participating site after trial rollout of eSyM. These patients were exposed to eSyM and used it to report symptoms.
Arm/Group | Cluster Randomized Trial (Intervention Patients - eSyM Responders) | Cluster Randomized Trial (Intervention Patients - eSyM Non-Responders)
Number analyzed (Participants) | 10078 | 10055
percentage of patients with event
  Medical Oncology: number analyzed (Participants) | 3593 | 4352
  Medical Oncology | 18.8 | 23.7
  Surgery: number analyzed (Participants) | 6485 | 5703
  Surgery | 10.8 | 16.1
  Medical Oncology + Surgery | 13.7 | 19.4
Statistical Analysis 1: Comparison: Cluster Randomized Trial (Intervention Patients - eSyM Responders) vs Cluster Randomized Trial (Intervention Patients - eSyM Non-Responders); [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 0.769, 95% CI 2-sided [0.729 to 0.811]
Statistical Analysis 2: Comparison: Cluster Randomized Trial (Intervention Patients - eSyM Responders) vs Cluster Randomized Trial (Intervention Patients - eSyM Non-Responders); Adjusted analysis comparing intervention responders versus non-responders (medical oncology patients only); Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 0.795, 95% CI 2-sided [0.737 to 0.858]
Statistical Analysis 3: Comparison: Cluster Randomized Trial (Intervention Patients - eSyM Responders) vs Cluster Randomized Trial (Intervention Patients - eSyM Non-Responders); Adjusted analysis comparing intervention responders versus non-responders (surgical patients only); Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 0.739, 95% CI 2-sided [0.686 to 0.796]

ADVERSE EVENTS:
Time Frame: Deaths during the study period were assessed for all trial patients for 1 year. Study-related adverse events were not monitored or collected during the study period because this intervention was deployed as a part of routine clinical care and the study was deemed minimal risk. All-cause mortality was evaluated as a study outcome.
Description: Since this was a research study deployed as a part of routine clinical care, formal adverse event reporting was not conducted.
Groups:
- eSyM Control Participants (Medical Oncology and Surgery Participants Combined): These patients (and/or proxy) were seen at a participating site prior to the trial rollout of eSyM and were not exposed to the eSyM intervention.
  This group includes the following trial subsets:
  * patients NOT exposed to the eSyM intervention through the stepped wedge cluster randomized trial (control cohort)
  * patients participating in the SASS control questionnaire
- eSyM Intervention Participants (Medical Oncology and Surgery Participants Combined): These patients (and/or proxy) were seen at a participating site after the trial rollout of eSyM and were exposed to the eSyM intervention.
  This group includes the following trial subsets:
  * patients exposed to the eSyM intervention through the stepped wedge cluster randomized trial (intervention cohort)
  * patients participating in the SASS intervention questionnaire
  * patients participating in qualitative interviews
  * patients participating in pilot testing
Arm/Group | eSyM Control Participants (Medical Oncology and Surgery Participants Combined) | eSyM Intervention Participants (Medical Oncology and Surgery Participants Combined)
All-Cause Mortality (participants affected / at risk) | 4898/21112 | 4161/18830
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-08-04): https://cdn.clinicaltrials.gov/large-docs/12/NCT03850912/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-12): https://cdn.clinicaltrials.gov/large-docs/12/NCT03850912/SAP_001.pdf